CLINICAL TRIAL: NCT02524548
Title: Improving Medication Adherence With Adjuvant Aromatase Inhibitor in Women With Breast Cancer: A Randomised Controlled Trial to Evaluate the Effect of Short Message Service (SMS) Reminder
Brief Title: SMS Reminders to Improve Medication Adherence of Aromatase Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Singapore Cancer Society (Other)
Responsible Party: Principal Investigator, Bee-Choo Tai, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DSRB 2014/01316
Record Dates: First submitted 2015-08-11; First posted 2015-08-17 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Medication Adherence
Keywords: Aromatase inhibitors; Reminder Systems
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS reminder (Experimental): Weekly SMS reminder to take aromatase inhibitors as prescribed by doctor
  Interventions: Other: SMS reminder
- Standard care (No Intervention): Routine care

INTERVENTIONS:
Other: SMS reminder — Weekly SMS reminder to take aromatase inhibitors as prescribed by doctor for 1 year
  Arms: SMS reminder

SUMMARY:
The purpose of this study is to determine whether weekly SMS reminders are effective in improving medication adherence of adjuvant aromatase inhibitors in women with breast cancer.

DETAILED DESCRIPTION:
This study is a prospective randomised controlled parallel trial of SMS reminder versus standard care to investigate whether SMS reminder improves adherence to oral aromatase inhibitor (AI) therapy amongst women with breast cancer at 1-year follow-up.

All subjects will be randomised to receive either SMS reminder or standard care in a 1:1 ratio. Balanced permuted block randomisation will be implemented with random varying of block sizes of 4 or 6.

The sample size is estimated based on the primary endpoint of medication adherence (as measured via SMAQ) at 1-year. Assuming that the proportion of medication adherence in the intervention and control groups are 80% and 60% respectively, then based on a 5% significance level and a power of 90%, a minimum sample of 240 subjects (i.e. 120 per group) will be required. Further assuming an attrition rate of 10%, the anticipated trial size is 280 overall.

The assessment of medication adherence at 1-year (as measured via SMAQ) between the SMS reminder and control groups will be made using chi-square test. Adjustment for baseline covariate and potential confounders will be made using the logistic regression where appropriate.

Other measures of adherence such as the 1-year MPR, PDC and pill count will be compared between treatment arms via the t- test, with adjustment for confounders made via the analysis of covariance (ANCOVA).

Natural log transformation will be implemented on the estrone and androstenedione measures to normalise the data. The assessment of secondary outcomes involving the log transformed estrone and androstenedione levels will be made using the analysis of covariance (ANCOVA) to adjust for the respective baseline levels and other potential confounders. Comparison of estradiol levels (defined as <18.4 versus ≥18.4) between the two arms will be made using chi-square test. The logistic regression analysis will be implemented to adjust for baseline covariate and other potential confounders where appropriate.

The assessment of knowledge, attitude, behavior, as well as barrier and facilitating factors between the intervention and control groups will be made using chi-square test, with treatment effect quantified based on odds ratio estimate and its 95% CI. Further adjustment for baseline scores and other potential confounders will be made using the logistic regression where appropriate.

Additionally, the investigators will compare the 4 different measures of adherence in a separate paper, to determine which of these provide a more meaningful or reliable information in the local context based on sensitivity analysis.

All analyses will be performed according to intention-to-treat using STATA, assuming a two-sided test at the 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have been receiving adjuvant endocrine therapy for at least 1 year, and are continuing to receive adjuvant AI therapy for at least 1 more year.
2. Have cellular phone that can receive text messages.
3. Singaporean or permanent resident who is currently residing in Singapore.
4. Able to give informed consent.

Exclusion Criteria:

1. Unable or not willing to comply with study procedures.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence | One year
  Simplified medication adherence questionnaire (SMAQ)

SECONDARY OUTCOMES:
Androstenedione | One year
  in nmol/L
Estrone | One year
  in pg/mL
Estradiol | One year
  in pmol/L

OTHER OUTCOMES:
Patients' knowledge, attitude, and behavior towards medication adherence | One year
  The Beliefs about Medicines Questionnaire (BMQ)
Patients' knowledge, attitude, and behavior towards medication adherence | One year
  Adherence Starts with Knowledge (ASK)-12 survey

CONTACTS AND LOCATIONS:
Overall Officials: Bee Choo Tai, PhD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He Y, Tan EH, Wong ALA, Tan CC, Wong P, Lee SC, Tai BC. Improving medication adherence with adjuvant aromatase inhibitor in women with breast cancer: study protocol of a randomised controlled trial to evaluate the effect of short message service (SMS) reminder. BMC Cancer. 2018 Jul 9;18(1):727. doi: 10.1186/s12885-018-4660-7. PMID 29986672